CLINICAL TRIAL: NCT03031470
Title: A Multicenter, Open-label, Randomized Pilot Clinical Study of Efficacy and Safety of Reparixin for Prevention of Early Allograft Dysfunction in Patients Undergoing Orthotopic Liver Transplantation
Brief Title: Pilot Study of Reparixin for Early Allograft Dysfunction Prevention in Liver Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Taking into account that 5 out of 22 patients in the Reparixin group experienced EAD during the first stage of the study, according to the Protocol and the DMC conclusion, it was decided on the early termination of the study
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPL-RPX-01
Record Dates: First submitted 2016-01-24; First posted 2017-01-25 (Estimated); Results first posted 2024-12-11 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Ischemia-reperfusion Injury in Liver Transplant; Early Allograft Dysfunction
Keywords: Liver Transplant; Ischemia-reperfusion injury; Early allograft dysfunction
MeSH Terms: conditions — Reperfusion Injury | interventions — reparixin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reparixin (Experimental): Patients in the group of the study therapy received Reparixin at dose of 2.772 mg/kg/hour for 7 days (168 hours). The prepared solution of Reparixin 11 mg/ml was administered as a continuous infusion into a central vein using an automatic infusion pump that provides a constant rate of infusion.
  All patients of the study received standard immunosuppressive therapy in accordance with the Russian Transplant Society Guidelines for liver transplantation.
  Interventions: Drug: Reparixin
- Control (Other): The patients, who were randomized in the control group, did not receive any study therapy. All patients of the study received standard immunosuppressive therapy in accordance with the Russian Transplant Society Guidelines for liver transplantation.
  Interventions: Other: Control

INTERVENTIONS:
Drug: Reparixin — Reparixin was administered as a continuous intravenous infusion for 7 days (Day 0 to Day 6) (168 hours).
  Reparixin was provided as 33 mg/ml concentrated solution to be diluted for i.v. infusion, packaged into 250 mL clear glass vials. To give a final concentration of 11 mg/mL, the content of a vial (250 ml) was diluted with 500 ml of 0.9% sterile saline to a total volume of 750 ml. The dosing solution was placed in a 1000 ml sterile empty Infusion Bag. Dosing solutions were to be used within 72 h from preparation, unless more restrictive rules.
  Reparixin infusion started approximately 60-90 minutes before the anticipated time of OLT. Infusion interruption was allowed for no more than 60 min.
  All patients received standard immunosuppressive therapy in accordance with the Russian Transplant Society Guidelines for liver transplantation.
  Patients and allograft survival were monitored up to 1 year after OLT.
  Arms: Reparixin
Other: Control — The patients who were randomized in the control group, did not receive any study therapy. The patients of both groups received the standard immunosuppressive therapy with Tacrolimus only or together with mycophenolates, or a combination of Tacrolimus/Cyclosporine with mycophenolates and/or glucocorticosteroids. The patients with hepatocellular carcinoma and impaired renal function could receive a combination of drugs that includes everolimus. Basiliximab in association with methylprednisolone was used for the induction of immunosuppression.
  Arms: Control

SUMMARY:
The objective of the study is to evaluate the efficacy and safety of Reparixin treatment (2.772 mg/kg body weight/hour intravenous continuous infusion for 7 days) based on incidence of early allograft dysfunction within the first 7 days after orthotopic liver transplantation (OLT) and overall indicators of allograft dysfunction in the early postoperative period (within 14 days after the OLT).

DETAILED DESCRIPTION:
The study is a phase 2, multicenter, open-label, randomized pilot study to evaluate the efficacy and safety of Reparixin for prevention of early allograft dysfunction in patients undergoing orthotopic liver transplantation.

All the patients who participated in the study received standard immunosuppressive therapy in accordance with the Russian Transplant Society Guidelines for liver transplantation (2013). The study was planned to be conducted at 5-8 transplantation sites in Russia and Belarus. Recruitment was competitive among the study sites so that patients were screened and if eligible, randomized consecutively until the randomization was stopped.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 years and older needing a whole organ OLT, listed on the waiting list for liver transplantation.
2. Severity score of the initial condition of the patient (hepatocellular dysfunction) according to the scales of Child-Turcotte-Pugh ≥ 7 points or MELD 15-40 points (or both).
3. The possibility of insertion of a central catheter for infusion of the study drug.
4. Signed Patient Informed Consent Form.
5. Ability to comply with all the requirements of the protocol.
6. Consent to use adequate contraception means throughout the study. The adequate contraception methods include use of condom with spermicide.

Exclusion Criteria:

Patients with any of the following conditions shall not be included in the study:

1. Split-liver transplantation or transplantation from a living donor.
2. Re-transplantation or multivisceral transplantation.
3. The presence of extrahepatic tumor foci or sepsis.
4. Gastrointestinal bleeding caused by portal hypertension within 3 months prior to screening.
5. BMI less than 18.5 or more than 40 kg/m2.
6. HIV infection.
7. Significant cardiovascular disease at the present time or within 6 months prior to screening, including: class III or IV chronic heart failure (the New York Heart Association), myocardial infarction, unstable angina, hemodynamically significant cardiac arrhythmias, ischemic or hemorrhagic stroke, uncontrolled arterial hypertension.
8. Preoperative renal impairment (glomerular filtration rate estimated with the Cockcroft-Gault formula ≤ 45 mL/min).
9. Significant, in the opinion of the Investigator, drug or alcohol abuse within 6 months prior to screening.
10. Hypersensitivity to:

    1. ibuprofen or to more than one non-steroidal anti-inflammatory drug (NSAID),
    2. more than one medication belonging to the class of sulfonamides, such as sulfamethazine, sulfamethoxazole, sulfasalazine, nimesulide or celecoxib; hypersensitivity to sulphanilamide antibiotics alone (e.g. sulfamethoxazole) does not qualify for exclusion.
11. Pregnant or lactating women, or women planning a pregnancy during the clinical study, fertile women not using adequate contraception methods.
12. Participation in another clinical study currently or within 30 days prior to screening, use of any investigational drug within 30 days or 5 half-lives (whichever is longer) prior to screening.
13. The patient's and his/her relatives' failure to understand the need for lifelong immunosuppressive therapy, as well as the risk and difficulty of the pending operation and the subsequent dynamic treatment.
14. Inability to read or write; unwillingness to understand and comply with the procedures of the study protocol; failure to comply with the treatment, which, in opinion of the Investigator, may affect the results of the study or the patient's safety and prevent the patient from further participation in the study; any other associated medical or serious mental conditions that make the patient unsuitable for participation in the clinical study, limit the validity of informed consent or may affect the patient's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03-10 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Vladimirovich Zhuravel, MD, Principal Investigator — Moscow Scientific Research Institute of Emergency, NV Sklifosovskiy of Moscow Healthcare Department
Locations (7):
- Healthcare Organization "9th City Clinical Hospital", Minsk, Belarus
- Russia (6):
  - State Budgetary Health Institution "Scientific Research Institute - Regional Clinical Hospital # 1 n.a. professor S.V. Ochapovskiy" of the Ministry of Health of the Krasnodar Territory, Krasnodar, Krasnodar Territory
  - State Budgetary Educational Institution of Higher Professional Education "First Saint Petersburg State Medical University n.a. I.P. Pavlov" of the Ministry of Health of the Russian Federation, Saint Petersburg, Sankt-Peterburg
  - Federal State Budgetary Institution "Academician V.I. Shumakov Federal Research Center of Transplantology and Artificial Organs" Ministry of Health of the Russian Federation, Moscow
  - Federal State Budgetary Institution "State Research Centre of the Russian Federation - Federal Medical Biophysical Centre n.a. A.I. Burnazyan", Moscow
  - State Budgetary Health Institution of Moscow "Scientific Research Institute of Emergency n.a. N.V. Sklifosovskiy of Moscow Healthcare Department", Moscow
  - State Budgetary Health Institution of Novosibirsk Region "State Novosibirsk Regional Clinical Hospital", Novosibirsk

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients admitted to the transplant center immediately before OLT surgery who signed the Patient Informed Consent Form underwent screening procedures (Day -1). Screening can be carried out within 24 hours before planned surgery. The results at screening were considered as baseline values.
  During the screening physical examination, patients fulfilling all the inclusion criteria and none of the exclusion criteria were randomized.
Groups:
- Reparixin: Patients in the group of the study therapy received Reparixin at dose of 2.772 mg/kg/hour for 7 days (168 hours). The prepared solution of Reparixin 11 mg/ml was administered as a continuous infusion into a central vein using an automatic infusion pump that provides a constant rate of infusion.
  Reparixin infusion started 60-90 minutes before OLT. Infusion interruption was allowed for no more than 60 minutes.
  All patients of the study received standard immunosuppressive therapy in accordance with the Russian Transplant Society Guidelines for liver transplantation.
  Reparixin: Reparixin was administered as a continuous intravenous infusion for 7 days (Day 0 to Day 6) (168 hours). Infusion of the study drug started approximately 60-90 minutes before the anticipated time of OLT (Orthotopic liver transplantation).The status of patients and allograft survival was monitored up to 1 year after OLT.
- Standard Care Procedures: The patients, who were randomized in the control group, did not receive any study therapy. All patients of the study received standard immunosuppressive therapy in accordance with the Russian Transplant Society Guidelines for liver transplantation.
  Standard care procedures: The patients, who were randomized in the control group, did not receive any study therapy. The patients of both groups received the standard immunosuppressive therapy with Tacrolimus only or together with mycophenolates, or a combination of Tacrolimus/Cyclosporine with mycophenolates and/or glucocorticosteroids. The patients with hepatocellular carcinoma and impaired renal function could receive a combination of drugs that includes everolimus. Basiliximab in association with methylprednisolone was used for the induction of immunosuppression.
Period: Overall Study
Arm/Group | Reparixin | Standard Care Procedures
Started | 22 | 18
Modified Intention to Treat Population (mITT) | 22 | 16
Per-Protocol Population (PP) | 17 | 16
Safety Population (SAF) | 22 | 16
Completed | 14 | 14
Not Completed | 8 | 4
Not completed — Adverse Event | 3 | 0
Not completed — Death | 3 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol entry criteria not met | 0 | 1
Not completed — Cancel the operation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified population of patients who received treatment (mITT = modified intent-to-treat) corresponds to all patients who received any dose of study drug. Two patients in the SoC arm didn't, so demographic characteristics of patients are listed for this population (n=22 in the Reparixin group and n=16 in the SoC group, for a total of n=38 patients instead of 40).
Groups:
- Reparixin - mITT: Patients in the group of the study therapy received Reparixin at dose of 2.772 mg/kg/hour for 7 days (168 hours). The prepared solution of Reparixin 11 mg/ml was administered as a continuous infusion into a central vein using an automatic infusion pump that provides a constant rate of infusion.
  Reparixin infusion started 60-90 minutes before OLT. Infusion interruption was allowed for no more than 60 minutes.
  All patients of the study received standard immunosuppressive therapy in accordance with the Russian Transplant Society Guidelines for liver transplantation.
  Reparixin: Reparixin was administered as a continuous intravenous infusion for 7 days (Day 0 to Day 6) (168 hours). Infusion of the study drug started approximately 60-90 minutes before the anticipated time of OLT (Orthotopic liver transplantation).The status of patients and allograft survival was monitored up to 1 year after OLT.
- Standard Care Procedures - mITT: The patients, who were randomized in the control group, did not receive any study therapy. All patients of the study received standard immunosuppressive therapy in accordance with the Russian Transplant Society Guidelines for liver transplantation.
  Standard care procedures: The patients, who were randomized in the control group, did not receive any study therapy. The patients of both groups received the standard immunosuppressive therapy with Tacrolimus only or together with mycophenolates, or a combination of Tacrolimus/Cyclosporine with mycophenolates and/or glucocorticosteroids. The patients with hepatocellular carcinoma and impaired renal function could receive a combination of drugs that includes everolimus. Basiliximab in association with methylprednisolone was used for the induction of immunosuppression.
- Total: Total of all reporting groups
Arm/Group | Reparixin - mITT | Standard Care Procedures - mITT | Total
Number analyzed (Participants) | 22 | 16 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 16 | 36
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (6.5) | 46.1 (9.5) | 50.7 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 11 | 29
  Male | 4 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 21 | 16 | 37
  Other - Mongoloid | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Belarus | 4 | 2 | 6
  Russia | 18 | 14 | 32

OUTCOME MEASURES:

1. Primary Outcome: Incidence of EAD (Early Allograft Dysfunction) Within 7 Days After OLT (PP Population)
Description: Assessment of the frequency of early allograft disfunction (EAD) after orthotopic liver transplantation (OLT) (Day 7 of Week 1) among patients who received Reparixin and patients in the control group. EAD was defined according to standard criteria as maximum Alanine Transferase (ALT) or Aspartate Transferase (AST) levels on days 1-7 of >2000 U/L, day 7 Bilirubin level ≥10 mg/dl, or a day 7 International Normalized ratio (INR) ≥1.6.
  Taking into account that 5 out of 22 patients in the Reparixin group experienced EAD during the first stage of the study, according to the Protocol and the DMC conclusion, it was decided on the early termination of the study.
Time Frame: within 7 day after the OLT
Population: Per protocol population (PP) includes all patients who have received at least 70% of the dose of the study drug, with data sufficient for the primary efficacy analysis, and who are considered compliant. Patients are considered compliant in case of absence of any major protocol violations during the study. In the group of the study therapy the patients who received not less than 70% of the study drug dose will be considered compliant.
Measure: Number (95% Confidence Interval); unit: percentage of participants with EAD
Groups:
- Reparixin - PP: Patients in the group of the study therapy received Reparixin at dose of 2.772 mg/kg/hour for 7 days (168 hours). The prepared solution of Reparixin 11 mg/ml was administered as a continuous infusion into a central vein using an automatic infusion pump that provides a constant rate of infusion.
  Reparixin infusion started 60-90 minutes before OLT. Infusion interruption was allowed for no more than 60 minutes.
  All patients of the study received standard immunosuppressive therapy in accordance with the Russian Transplant Society Guidelines for liver transplantation.
  Reparixin: Reparixin was administered as a continuous intravenous infusion for 7 days (Day 0 to Day 6) (168 hours). Infusion of the study drug started approximately 60-90 minutes before the anticipated time of OLT (Orthotopic liver transplantation).The status of patients and allograft survival was monitored up to 1 year after OLT.
- Control - PP: The patients, who were randomized in the control group, did not receive any study therapy. All patients of the study received standard immunosuppressive therapy in accordance with the Russian Transplant Society Guidelines for liver transplantation.
  Control: The patients, who were randomized in the control group, did not receive any study therapy. The patients of both groups received the standard immunosuppressive therapy with Tacrolimus only or together with mycophenolates, or a combination of Tacrolimus/Cyclosporine with mycophenolates and/or glucocorticosteroids. The patients with hepatocellular carcinoma and impaired renal function could receive a combination of drugs that includes everolimus. Basiliximab in association with methylprednisolone was used for the induction of immunosuppression.
Arm/Group | Reparixin - PP | Control - PP
Number analyzed (Participants) | 17 | 16
percentage of participants with EAD | 29.4 [10.3 to 56.0] | 18.8 [4.0 to 45.6]
Statistical Analysis 1: Comparison: Reparixin - PP vs Control - PP; Test type: Superiority; p = 0.688, Fisher Exact; Analysis is based on exact Fisher test to compare treatments

2. Primary Outcome: Incidence of EAD (Early Allograft Dysfunction) Within 7 Days After OLT (mITT Population)
Description: Assessment of the frequency of early allograft disfunction after orthotopic liver transplantation (OLT) (Day 7 of Week 1) among patients who received Reparixin and patients in the control group. EAD was defined according to standard criteria as maximum Alanine Transferase (ALT) or Aspartate Transferase (AST) levels on days 1-7 of >2000 U/L, day 7 Bilirubin level ≥10 mg/dl, or a day 7 International Normalized ratio (INR) ≥1.6.
  Please note that taking into account that 5 out of 22 patients in the Reparixin group experienced EAD during the first stage of the study, according to the Protocol and the DMC conclusion, it was decided on the early termination of the study.
Time Frame: within 7 day after the OLT
Population: Modified population of patients who received treatment (MITT = modified intent-to-treat) corresponds to all patients who received any dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants with EAD
Groups:
- Control - mITT: The patients, who were randomized in the control group, did not receive any study therapy. All patients of the study received standard immunosuppressive therapy in accordance with the Russian Transplant Society Guidelines for liver transplantation.
  Control: The patients, who were randomized in the control group, did not receive any study therapy. The patients of both groups received the standard immunosuppressive therapy with Tacrolimus only or together with mycophenolates, or a combination of Tacrolimus/Cyclosporine with mycophenolates and/or glucocorticosteroids. The patients with hepatocellular carcinoma and impaired renal function could receive a combination of drugs that includes everolimus. Basiliximab in association with methylprednisolone was used for the induction of immunosuppression.
Arm/Group | Reparixin - mITT | Control - mITT
Number analyzed (Participants) | 22 | 16
percentage of participants with EAD | 22.7 [9.1 to 51.2] | 18.8 [4.0 to 45.6]
Statistical Analysis 1: Comparison: Reparixin - mITT vs Control - mITT; Test type: Superiority; p = 0.700, Fisher Exact; Analysis is based on exact Fisher test to compare treatments

3. Secondary Outcome: Number of Patients With/Without Primary Allograft Nonfunction Within 7 Days After OLT
Description: The number of patients in which: a) the primary allograft nonfunction within 7 day after the OLT was determined and not determined, and the number of patients in which 2)Appropriate data was not available in each of the two arms are reported.
Time Frame: Within 7 days after OLT
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Reparixin - mITT | Standard Care Procedures - mITT
Number analyzed (Participants) | 22 | 16
Participants
  Primary nonfunction - No | 17 | 12
  Primary nonfunction - yes | 0 | 0
  No data | 5 | 4
Statistical Analysis 1: Comparison: Reparixin - mITT vs Standard Care Procedures - mITT; Test type: Superiority; p > 0.999, Fisher Exact; Treatment groups were compared for frequency of allograft nonfunction using Fisher exact test

4. Secondary Outcome: Number of Patients With/Without Overall Indicators of Allograft Dysfunction During the Early Postoperative Period
Description: The number of patients in which: a) the primary allograft dysfunction within 14 day after the OLT was determined and not determined, and the number of patients in which 2)Appropriate data was not available in each of the two arms are reported. The term "early allograft dysfunction" (EAD) identifies liver transplant (LT) allografts with initial poor function and portends poor allograft and patient survival.
Time Frame: Within 14 days after OLT
Population: as for outcome 2
Measure: Number; unit: participants with allograft dysfunction
Arm/Group | Reparixin | Standard Care Procedures
Number analyzed (Participants) | 22 | 16
participants with allograft dysfunction
  yes | 5 | 3
  no | 14 | 13
  No data | 3 | 0
Statistical Analysis 1: Comparison: Reparixin vs Standard Care Procedures; Test type: Superiority; p = 0.308, Fisher Exact

5. Secondary Outcome: Overall Indicators of the Allograft Dysfunction During the Early Postoperative Period - Extracorporeal Detoxification
Description: Cumulative incidence of extracorporeal detoxification as an indicator of liver allograft dysfunction in early postoperative period within 2 weeks after OLT is reported. Extracorporeal liver support describes all measures of extracorporeal blood treatments, which are aimed at supporting any functions of the liver in order to reduce the number of failing organs as a consequence of liver failure. The ultimate goal of extracorporeal liver support is to prolong the survival time of patients with liver failure by preventing progression of secondary organ failure.
Time Frame: Within 14 days after OLT
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Reparixin - mITT | Standard Care Procedures - mITT
Number analyzed (Participants) | 22 | 16
Participants | 0 | 0
Statistical Analysis 1: Comparison: Reparixin - mITT vs Standard Care Procedures - mITT; Test type: Superiority; p = 0.601, Fisher Exact

6. Secondary Outcome: Frequency of Identification of Laboratory Examination Values
Description: The frequency of identification of laboratory examination values corresponding to early allograft dysfunction within 3 days after the operation (Day 4 of the study drug administration)
Time Frame: within 3 day after the OLT
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Reparixin - mITT | Standard Care Procedures - mITT
Number analyzed (Participants) | 22 | 16
Participants
  ALT> 2000 U/L | 1 | 0
  AST> 2000 U/L | 0 | 0
  AST and ALT > 2000 U/L | 0 | 0

7. Secondary Outcome: Number of Patients With Early Allograft Dysfunction (EAD) in Case of Transplantation of Donor Organs, by the Degree of Steatosis
Description: Incidence of early allograft dysfunction in case of transplantation of donor organs differing by the degree of steatosis was reported.
  The investigators evaluated organ suitability for transplantation relying on histopathologic findings from biopsy. In this clinical setting, grafts with macrovesicular steatosis degree >50% were considered as non-suitable for transplantation.
  Steatosis or fatty liver disease (NAFLD) is characterised by hepatic lipid accumulation. Nominal data for the MITT are reported.
Time Frame: Within 14 days after OLT
Population: as for outcome 2
Measure: Number; unit: Subjects with EAD
Arm/Group | Reparixin - mITT | Standard Care Procedures - mITT
Number analyzed (Participants) | 22 | 16
Subjects with EAD
  participants with allograft steatosis within 0 - 10 % | 0 | 2
  participants with allograft steatosis within 10 - 30 % | 5 | 1
  participants with allograft steatosis within 30 - 50 % | 0 | 0
Statistical Analysis 1: Comparison: Reparixin - mITT vs Standard Care Procedures - mITT; Test type: Superiority; p = 0.574, Cochran-Mantel-Haenszel; Reparixin and Control groups will be compared for degree of allograft steatosis using Cochran-Mantel-Hensel (CMH) test with control EAD

8. Secondary Outcome: Number of Patients With EAD in Case of Transplantation of Donor Organs Differing by the Time (in Hours) of Allograft Removal From the Donor and up to Its Reperfusion (Duration of Cold Ischemia)
Description: Number of patients with EAD in case of transplantation of donor organs by the time of allograft removal from the donor and up to its reperfusion after engraftment (duration of cold ischemia) was assessed.
  Cold ischemia time during procurement is defined as the time after clamping of aorta until excision of the organ, which can last some hours. Prolonged cold ischemia time is an independent risk factor for the development of delayed function and primary nonfunction of the allograft. Although the exact mechanism is unknown, cold ischemia time is believed to affect graft function by contributing to ischemia-reperfusion injury. Nominal data for the MITT are reported.
Time Frame: Within 14 days after OLT
Population: as for outcome 2
Measure: Number; unit: number of participants
Arm/Group | Reparixin - mITT | Standard Care Procedures - mITT
Number analyzed (Participants) | 22 | 16
number of participants
  patients who had a duration of cold ischemia < 5 hours | 0 | 1
  patients who had a duration of cold ischemia of 5-6 hours | 0 | 1
  patients who had a duration of cold ischemia of 6-7 hours | 4 | 1
  patients who had a duration of cold ischemia of more than 7 hours | 1 | 0
Statistical Analysis 1: Comparison: Reparixin - mITT vs Standard Care Procedures - mITT; Test type: Superiority; p = 0.843, Cochran-Mantel-Haenszel; Reparixin and Control groups will be compared for duration of cold ischemia using Cochran-Mantel-Hensel (CMH) test with control EAD

9. Secondary Outcome: Number of Patients With EAD in Case of Transplantation of Donor Organs Differing by the Duration (in Min) of Warm Ischemia
Description: The number of EAD patients in case of transplantation of donor organs differing by the time of allograft removal from the donor and up to its reperfusion after engraftment (duration of warm ischemia) was assessed. In surgery, warm ischemia is the time a tissue, organ, or body part remains at body temperature after its blood supply has been reduced or cut off but before it is cooled or reconnected to a blood supply. In the transplant setting, this term is used to describe two physiologically distinct periods of ischaemia: (1) Ischemia during implantation, from removal of the organ from ice until reperfusion, and (2) Ischemia during organ retrieval, from the time of cross clamping (or of asystole in non-heart-beating donors), until cold perfusion is commenced. Nominal data for the MITT are reported.
Time Frame: Within 14 days after OLT
Population: Modified population of patients who received treatment (mITT = modified intent-to-treat) corresponds to all patients who received any dose of study drug. While 3 patients in the SoC are reported to develop EAD, data regarding the duration of warm ischemia are available for only 2 patients in the SoC arm.
Measure: Number; unit: number of participants
Arm/Group | Reparixin - mITT | Standard Care Procedures - mITT
Number analyzed (Participants) | 22 | 16
number of participants
  patients who had a duration of warm ischemia < 30 minutes | 1 | 0
  patients who had a duration of warm ischemia of 30 - 45 minutes | 3 | 1
  patients who had a duration of warm ischemia of 46 - 60 minutes | 0 | 1
  patients who had a duration of warm ischemia > 60 minutes | 0 | 0
Statistical Analysis 1: Comparison: Reparixin - mITT vs Standard Care Procedures - mITT; Test type: Superiority; p = 0.701, Cochran-Mantel-Haenszel; Reparixin and Control groups will be compared for duration of earm ischemia using Cochran-Mantel-Hensel (CMH) test with control EAD

10. Secondary Outcome: Number of Patients With EAD in Transplantation From Donors Having Additional Adverse Factors
Description: The number of patients with early allograft dysfunction in transplantation from donors having additional adverse factors like infectious complication, death of the brain, hypotension, etc. was reported. The correlation between EAD and additional adverse factors are showed. Nominal data for the MITT are reported.
Time Frame: Within 14 days after OLT
Population: as for outcome 2
Measure: Number; unit: patients with additional adverse fact
Arm/Group | Reparixin - mITT | Standard Care Procedures - mITT
Number analyzed (Participants) | 22 | 16
patients with additional adverse fact
  Infectious complications -yes | 0 | 0
  Death of the brain -yes | 5 | 3
  Hypotension - yes | 0 | 0
  Other - yes | 0 | 0

11. Secondary Outcome: Number of Patients With EAD in Transplantation With Regard to the Interval (in Hours) Between the Diagnosis of Brain Death and Removal of the Liver Graft From a Donor
Description: The number of patients with allograft dysfunction in transplantation with regard to the interval between the diagnosis of brain death and removal of the liver graft from a donor (in the case of a brain-dead donor). This interval can last hours. Nominal data for the mITT are reported.
Time Frame: Within 14 days after OLT
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Reparixin - mITT | Standard Care Procedures - mITT
Number analyzed (Participants) | 22 | 16
participants
  less than 2 hours | 1 | 0
  2,3 hours | 0 | 1
  3,4 hours | 1 | 1
  4,6 hours | 2 | 0
  6,8 hours | 0 | 0
  more than 8 hours | 1 | 1

12. Secondary Outcome: Number of Patients With EAD in Transplant Recipients With Each of the Different Liver Disease Etiology
Description: The number of patients with EAD in transplant recipients with liver diseases of different etiology (viral, alcoholic, autoimmune, etc.) was assessed.
Time Frame: Within 14 days after OLT
Population: as for outcome 2
Measure: Number; unit: participants with liver diseases
Units Other Than Participants: early allograft dysfunction detected
Arm/Group | Reparixin - mITT | Standard Care Procedures - mITT
Number analyzed (Participants) | 22 | 16
Number analyzed (early allograft dysfunction detected) | 5 | 3
participants with liver diseases
  recipients with Viral disease etiology - yes | 2 | 3
  recipients with Alcoholic disease etiology - yes | 1 | 0
  recipients with Autoimmune disease etiology - yes | 1 | 0
  recipients with other disease etiology - Cirrhosis HCV + HCC in segment VII or Cryptogenic or toxic | 1 | 0

13. Secondary Outcome: Incidence of Early Allograft Dysfunction (EAD) in Transplant Recipients With Liver Diseases of Different Etiology and With Different Baseline Characteristics
Description: The incidence of early allograft dysfunction in transplant recipients with liver diseases of different etiology and with different baseline characteristics.
  Herein the intent is reporting the number/percentage of subjects with EAD within 14 days after OLT, without distinction for disease etiology and baseline characteristics.
Time Frame: Within 14 days after OLT
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Reparixin - mITT | Standard Care Procedures - mITT
Number analyzed (Participants) | 22 | 16
Participants | 5 | 3

14. Secondary Outcome: The Number of Patients With EAD in Transplant Recipients With Liver Diseases (HBV and HCV Virus) and With Different Baseline Characteristics
Description: The number of EAD patients in transplant recipients with liver diseases detected, and with different baseline characteristics was assessed. Herein HBV and HCV viral load at screening visit are reported.
Time Frame: Within 14 days after OLT
Population: as for outcome 2
Measure: Number; unit: participants with viral load
Arm/Group | Reparixin - mITT | Standard Care Procedures - mITT
Number analyzed (Participants) | 22 | 16
participants with viral load
  HBV virus loading - detected | 0 | 0
  HBV virus loading - not detected | 3 | 2
  HCV virus loading - detected | 1 | 1
  HCV virus loading - not detected | 2 | 2

15. Secondary Outcome: Incidence of Early Allograft Dysfunction in Transplant Recipients (Creatinine Clearance, ClCr)
Description: The incidence of early allograft dysfunction in transplant recipients with different baseline characteristics. Herein Creatinine clearance at screening Day - 1 (mL/min). Creatinine clearance (CrCl) is the volume of blood plasma cleared of creatinine per unit time. It is a rapid and cost-effective method for the measurement of renal function. the normal range of CrCl is 110 to 150mL/min in males and 100 to 130mL/min in females. Serum creatinine level for men with normal kidney function is approximately 0.6 to 1.2mg/dL and between 0.5 to 1.1 mg/dL for women. Creatine levels above the normal range indicate renal dysfunction.
Time Frame: Within 14 days after OLT
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Reparixin - mITT | Standard Care Procedures - mITT
Number analyzed (Participants) | 22 | 16
ml/min | 81.6 (30.1) | 73.5 (20.0)

16. Secondary Outcome: Incidence of Early Allograft Dysfunction in Transplant Recipients - Severity of Recipient's Liver Disease Through MELD Index
Description: The incidence of early allograft dysfunction in transplant recipients with different score in scales of end-stage liver disease. The MELD score estimates a patient's chances of surviving their disease during the next three months. Practically, MELD is a reliable measure of mortality risk in patients with end-stage liver disease. It is used as a disease severity index to determine prognosis and help prioritize patients for organ allocation by estimating 3-month mortality risk. The MELD score ranges from 6 to 40 and is based on results from several lab tests. The higher the number, the more likely the subject is to receive a liver from a deceased donor when an organ becomes available.
  MELD Score= 11.2 x In INR + 9.57 x In Creatinine (mg/dL) + 3.78 (if the patient had dialysis at least twice in the past week, the value for serum creatinine needs to be adjusted to 4.0) x In Bilirubine (mg/dL) + 6.43
Time Frame: Within 14 days after OLT
Population: as for outcome 2
Measure: Number; unit: recipients with liver disease via MELD
Arm/Group | Reparixin - mITT | Standard Care Procedures - mITT
Number analyzed (Participants) | 22 | 16
recipients with liver disease via MELD
  < 9 - 1.9% mortality | 0 | 0
  10 - 19 - 6.0% mortality | 5 | 2
  20 - 29 - 19.6% mortality | 0 | 1
  30 - 39 - 52.6% mortality | 0 | 0

17. Secondary Outcome: Number of Patients With EAD in Transplant Recipients Via Child-Turcotte-Pugh Score (CTP)
Description: The incidence of early allograft dysfunction in transplant recipients with different allograft dysfunction based on CTP. This score assesses the severity of the disease, the risk of lethal outcome (during surgeries) and the prognosis in patients with cirrhosis. The CTP scoring system incorporates five parameters: serum bilirubin, serum albumin, prothrombin time, ascites, and grade of encephalopathy.
  Each of them can score between 1 and 3. Based on the sum of the points from these five parameters, the patient is categorized into one of three CTP classes/grades: A, B, or C.
  Score:
  • 5-6 points - Grade A (least severe liver disease)
  * 7-9 points - Grade B (moderately severe liver disease)
  * 10-15 points - Grade C (most severe liver disease)
Time Frame: Within 14 days after OLT
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Reparixin - mITT | Standard Care Procedures - mITT
Number analyzed (Participants) | 22 | 16
participants
  5-6 points Grade А (least severe liver disease) | 0 | 0
  7-9 points Grade В (moderately severe liver disease) | 4 | 1
  10-15 points Grade С (most severe liver disease) | 1 | 2

18. Secondary Outcome: Time to Liver Function Normalization of Liver Function Parameters
Description: Time to normalization of liver function parameters (alanine aminotransferase, aspartate aminotransferase and bilirubin levels, gamma-glutamyltransferase, lactate dehydrogenase, etc.) after the OLT was assessed. Please note the upper limit of IC is not available due to insufficient number of participants with events.
Time Frame: Within 1 Year after OLT
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Reparixin - mITT | Standard Care Procedures - mITT
Number analyzed (Participants) | 22 | 16
hours | 87 [84 to NA] — Upper 95% CI confidence interval value was not achieved due to insufficient number of observations. | NA [NA to NA] — Median with 95% CI for the time from the OLT to normalization of liver parameters was not achieved for patients in the Control group due to insufficient number of observations.

19. Secondary Outcome: Patient Survival Within 1 Year After OLT
Description: Patient survival within 1 year after OLT was assessed. Please note the data are not available due to insufficient number of participants with events.
Time Frame: within 1 year after OLT
Population: Modified population of patients who received treatment (mITT = modified intent-to-treat) corresponds to all patients who received any dose of study drug. Please note data are not available due to insufficient number of participants with events.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Reparixin - mITT | Standard Care Procedures - mITT
Number analyzed (Participants) | 22 | 16
days | NA [NA to NA] — Survival Kaplan-Mayer curve shows that median survival time could not be measured. | NA [NA to NA] — Survival Kaplan-Mayer curve shows that median survival time could not be measured.
Statistical Analysis 1: Comparison: Reparixin - mITT vs Standard Care Procedures - mITT; Test type: Superiority — General survival and graft survival ("graft loss" will be qualified as an event for "graft survival") within 1 year were presented with Kaplan-Mayer curves and survival time median with 95% CI. Treatment groups will be compared using logrank test; p = 0.416, Log Rank

20. Secondary Outcome: Mortality Within 1 Year After the OLT
Description: Number of deaths within 1 year after the OLT was assessed.
Time Frame: Within 1 Year after OLT
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Reparixin - mITT | Control - mITT
Number analyzed (Participants) | 22 | 16
Participants | 4 | 1

21. Secondary Outcome: The Incidence of Hyperacute, Acute and Chronic Liver Allograft Rejection .
Description: Hyperacute or acute transplant rejection were determined by biopsy; chronic transplant rejection was defined by histological evaluation in both treatment groups.
Time Frame: Within 1 Year after OLT
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Reparixin - mITT | Control - mITT
Number analyzed (Participants) | 22 | 16
participants
  hyperacute | 0 | 0
  acute | 0 | 0
  chronic | 0 | 0

22. Secondary Outcome: Summary of Adverse Events up to 1 Year After the OLT
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign (including abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: up to 1 year after the OLT
Population: SAF= Set of patients called the Safety population; patients are grouped for analysis according to the treatment they actually received, as opposed to the treatment they were allocated to receive at randomization.
Measure: Number; unit: participants with AE
Groups:
- Control: The patients, who were randomized in the control group, did not receive any study therapy. All patients of the study received standard immunosuppressive therapy in accordance with the Russian Transplant Society Guidelines for liver transplantation.
  Control: The patients, who were randomized in the control group, did not receive any study therapy. The patients of both groups received the standard immunosuppressive therapy with Tacrolimus only or together with mycophenolates, or a combination of Tacrolimus/Cyclosporine with mycophenolates and/or glucocorticosteroids. The patients with hepatocellular carcinoma and impaired renal function could receive a combination of drugs that includes everolimus. Basiliximab in association with methylprednisolone was used for the induction of immunosuppression.
Arm/Group | Reparixin | Control
Number analyzed (Participants) | 22 | 16
participants with AE
  Number (%) of patients reporting at least one AE | 20 | 13
  Number (%) of patients reporting at least one AE leading to discontinuation of study drug | 3 | 0
  Number (%) of patients reporting at least one serious AE | 16 | 5

ADVERSE EVENTS:
Time Frame: The specific period of time over wich adverse events data were collected was up to 12 weeks after the OLT and 1 year after OLT. Herein the summary of Adverse Events up to 1 year after OLT was reported.
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign (including abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Groups:
- Reparixin - SAF: Patients in the group of the study therapy received Reparixin at dose of 2.772 mg/kg/hour for 7 days (168 hours). The prepared solution of Reparixin 11 mg/ml was administered as a continuous infusion into a central vein using an automatic infusion pump that provides a constant rate of infusion.
  Reparixin infusion started 60-90 minutes before OLT. Infusion interruption was allowed for no more than 60 minutes.
  All patients of the study received standard immunosuppressive therapy in accordance with the Russian Transplant Society Guidelines for liver transplantation.
  Reparixin: Reparixin was administered as a continuous intravenous infusion for 7 days (Day 0 to Day 6) (168 hours). Infusion of the study drug started approximately 60-90 minutes before the anticipated time of OLT (Orthotopic liver transplantation).The status of patients and allograft survival was monitored up to 1 year after OLT.
- Standard Care Procedures - SAF: The patients, who were randomized in the control group, did not receive any study therapy. All patients of the study received standard immunosuppressive therapy in accordance with the Russian Transplant Society Guidelines for liver transplantation.
  Standard care procedures: The patients, who were randomized in the control group, did not receive any study therapy. The patients of both groups received the standard immunosuppressive therapy with Tacrolimus only or together with mycophenolates, or a combination of Tacrolimus/Cyclosporine with mycophenolates and/or glucocorticosteroids. The patients with hepatocellular carcinoma and impaired renal function could receive a combination of drugs that includes everolimus. Basiliximab in association with methylprednisolone was used for the induction of immunosuppression.
Arm/Group | Reparixin - SAF | Standard Care Procedures - SAF
All-Cause Mortality (participants affected / at risk) | 4/22 | 1/16
Serious Adverse Events (participants affected / at risk) | 16/22 | 5/16
Other Adverse Events (participants affected / at risk) | 20/22 | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reparixin - SAF (N=22) | Standard Care Procedures - SAF (N=16)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hernial eventration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus spastic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary ischaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic artery thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver transplant rejection (Immune system disorders) | 0 (0) | 1 (1)
Transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Chemical peritonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Complications of transplanted liver (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reparixin - SAF (N=22) | Standard Care Procedures - SAF (N=16)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 4 (6)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 3 (4) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 2 (3)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Biliary ischaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal vein stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 2 (2) | 1 (1)
Hepatitis B (Infections and infestations) | 2 (2) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (2) | 3 (4)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 4 (4)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Viraemia (Infections and infestations) | 0 (0) | 1 (1)
Wound abscess (Infections and infestations) | 1 (1) | 0 (0)
Anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Complications of transplanted liver (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative hernia (Infections and infestations) | 3 (3) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suture rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transplant dysfunction (Injury, poisoning and procedural complications) | 5 (5) | 2 (3)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 2 (2) | 2 (2)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (3) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 7 (7)
Haematoma (Vascular disorders) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Post thrombotic syndrome (Vascular disorders) | 1 (1) | 0 (0)
Hernial eventration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-03-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT03031470/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/70/NCT03031470/SAP_001.pdf